CLINICAL TRIAL: NCT05385874
Title: Risk Prediction and Its Intelligent Assessment for Cognitive Impairment Among Community-dwelling Older Adults
Status: Completed | Type: Observational
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xiaozhen LV, Associate Researcher, Peking University Sixth Hospital
Other Study IDs: SHOUFA2020-3-4114
Record Dates: First submitted 2022-05-11; First posted 2022-05-23 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Impairment; Predictive Model; Aging; Cohort
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: The training cohort will be used for model development.
- Testing cohort: The testing cohort, a new cohort compared with the training cohort, will be used for model external validation.

SUMMARY:
Cognitive impairment is one of the core early signs of dementia, and it is also a key stage for community-based dementia prevention. Accurate and convenient prediction of cognitive impairment can help the community to identify and manage the high-risk population of dementia. Previous studies had developed several dementia predicting models, but such models may be not suitable for cognitive impairment prediction. Based on the national representative follow-up data of Chinese Longitudinal Healthy Longevity Survey (CLHLS), this project aims to develop and validate a brief cognitive impairment prediction algorithm among the community-dwelling elderly, using machine learning methods (such as Logistic regression, Naïve Bayes model, Extreme Gradient Boosting Tree and so on). Finally, based on the constructed model, an easy-to-use online intelligent assessment tool for predicting cognitive impairment risk will be developed. The general practitioners, social workers and the elderly would be invited to use the tool and we will revise the tool according to their suggestions and comments. This project is expected to provide scientific basis and technical support for community-based dementia prevention, and will also be useful for the elderly to easily understand their cognitive health.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or over at baseline;
2. With normal cognitive function at baseline (score ≥ 18 on the Chinese version of Mini-Mental State Examination, MMSE);
3. Completed MMSE assessment three years later;
4. Provided informed consent voluntarily.

Exclusion Criteria:

1. Aged <65;
2. had a history of dementia or MMSE score < 18 at baseline;
3. lost to follow-up or without cognitive function assessment three years later;
4. Refused to participate the survey.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population of this project was those community-dwelling older adults with normal cognitive function at baseline and completed cognitive function assessment three years later.
Sampling Method: Non-Probability Sample
Enrollment: 13228 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
AUC | an average of 3 years after baseline assessement
  the AUC of the prediciton model based on the test data

SECONDARY OUTCOMES:
sensitivity | an average of 3 years after baseline assessement
  the sensitivity of the prediciton model based on the test data
specificity | an average of 3 years after baseline assessement
  the specificity of the prediciton model based on the test data
positive predictive value | an average of 3 years after baseline assessement
  the positive predictive value of the prediciton model based on the test data
negative predictive value | an average of 3 years after baseline assessement
  the negative predictive value of the prediciton model based on the test data

CONTACTS AND LOCATIONS:
Overall Officials: Feifei Gao, Ph.D, Study Director — Peking University Six Hospital
Locations (1):
- Peking University Six Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided